CLINICAL TRIAL: NCT05171673
Title: A Multi-center, Prospective, Open-label, Controlled Study of the Pharmacokinetics and Safety of the LicartTM Topical System in Pediatric and Adult Participants with Minor Soft Tissue Injuries
Brief Title: Study of PK and Safety of the LicartTM Topical System in Pediatric and Adult Participants with Minor Soft Tissue Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18US-FHp04
Record Dates: First submitted 2021-11-09; First posted 2021-12-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Soft Tissue Injuries
MeSH Terms: conditions — Soft Tissue Injuries | interventions — diclofenac hydroxyethylpyrrolidine; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Open-label, controlled study in pediatric and adult participants with minor soft tissue injuries. One-hundred fifty (150) participants between 6 and 11years old; 12 and 16 years old; and 18 and 45 years old will be enrolled, with equal numbers in each of the three age groups. The 50 adults enrolled will serve as the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational (Experimental): LicartTM topical system application once per day for a maximum of 14 days or until pain resolution, whichever occurs first.
  Interventions: Drug: Licart™ (diclofenac epolamine) topical system

INTERVENTIONS:
Drug: Licart™ (diclofenac epolamine) topical system — The Licart™ (diclofenac epolamine) topical system was designed to deliver the nonsteroidal anti-inflammatory drug (NSAID) diclofenac to the site of a minor soft tissue injury through topical application. This investigational product (IP) is a 10 cm x 14 cm topical system comprised of an adhesive material containing 1.3% diclofenac epolamine that is bound to a non-woven polyester felt backing and covered with a polypropylene film release liner. The release liner is removed prior to topical application to the skin.
  Other Names: diclofenac epolamine

SUMMARY:
A multi-center, prospective, open-label, controlled study of the pharmacokinetics and safety of the LicartTM topical system in pediatric and adult participants with minor soft tissue injuries. 150 male and female participants aged 6-16 and 18-45 with soft tissue injuries meeting the following criteria will be enrolled to evaluate the pharmacokinetics and safety of the Licart topical system in pediatric and adult participants with minor soft tissue injuries over a 14-day treatment course. The analgesic effects will also be evaluated of the topical system in pediatric and adult participants with minor soft tissue injuries over a 14-day treatment course. To collect principal investigator-reported global response to therapy.

DETAILED DESCRIPTION:
Open-label, controlled study in pediatric and adult participants with minor soft tissue injuries. One-hundred fifty (150) participants between 6 and 11years old; 12 and 16 years old; and 18 and 45 years old will be enrolled, with equal numbers in each of the three age groups. The 50 adults enrolled will serve as the control. Participants will be seen by the principal investigator (PI) or designee at the clinical site, at entry and Visits 2 and 5 following the first topical system application, with the last visit scheduled on either Day 14 or the day after the participant experiences pain resolution. Visits 3 and 4 will be conducted via telehealth. At each study visit, adverse events (AEs) and concomitant medications will be recorded, local tolerability at the application site scored on a 7-point scale, and pain assessed by participants using the Wong-Baker FACES scale. Vital signs will be measured at the screening visit and Visits 2 and 5.

Participants will also assess pain twice daily (morning and evening) at home in the Participant Diary using the same Wong-Baker FACES scale. Blood samples will be obtained from each participant at Visit 2, 24 hours (± 1 hour) after initial topical system application at Visit 1, and at the time of study discontinuation (with a topical system in place) for determination of plasma diclofenac concentration and plasma activated partial thromboplastin time (aPTT). At the End-of-Study (EOS) Visit the principal investigator will provide an assessment of global response to therapy on a 5-point scale.

Participants will be asked to apply the Licart topical system once per day for a maximum of 14 days or until pain resolution, whichever occurs first.

This study will assess efficacy by the following assessments: Plasma diclofenac concentration, 24 hours (± 1 hour) after initial application (Visit 2) and EOS Visit; Pain score assessment by participant using the Wong-Baker FACES scale: every day (Participant Diary) and study visits on Visits 2, 3, 4 and 5; and Principal investigator assessment of global response to therapy on a 5-point scale.

This study will assess safety by the following assessments: Vital signs will be measured at the screening visit and Visit 2 and 5; AE reporting at each study visit; Local tolerability on a 7-point scale at Visits 2, 3, 4 and 5, or the day after pain resolution, with a topical system applied to the injured area; Plasma diclofenac concentration, 24 hours (±1 hour) after initial topical system application (Visit 2) and EOS Visit; and Plasma activated partial thromboplastin time (aPTT), 24 hours (±1 hour) after initial topical system application (Visit 2) and EOS Visit.

The primary endpoints of the study are: Diclofenac pharmacokinetic profile (Pediatric population vs Adult population; Two-sided 90% confidence interval (CI) <4 ng/mL); Local tolerability; AEs; and Activated partial thromboplastin time (aPTT).

The secondary endpoints of the study are: Participant-reported pain scores; Global response to therapy; and Vital signs.

All participants who receive at least one topical system will be subjected to classic safety and efficacy analyses. All participants who receive at least one topical system and have at least one blood draw to support determination of plasma diclofenac concentration will be subjected to the pharmacokinetic analysis. An evaluable participant population with adequate compliance and follow- up may also be analyzed.

Continuous variables will be presented as sample size, means, medians, standard deviations, range and 90% CI. Categorical variables will be presented as sample size, number of observations, percentages and exact 90% CI.

The participant population will be stratified by appropriate age categories and the effects of age may be analyzed using Analysis of Variance (ANOVA) or multiple regression methods.

Plasma diclofenac concentration in pediatric participants will be compared with those of adults using repeated measures mixed models (participants will have reached steady-state blood concentration by the time of the first blood draw).

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent;
2. Male or female, 6-11 years old; 12-16 years old; or 18-45 years old;
3. BMI <32kg/m2;
4. Minor soft tissue injury within 96 hours of enrollment;
5. Spontaneous pain of at least moderate intensity (i.e., pain of at least 6 on the Wong-Baker FACES® scale) according to the participant);
6. Clinically significant injury according to the principal investigator;
7. Willing and able to accommodate study requirements for data collection, including return for study Visits 2 and 5;
8. Have access to high-speed internet, a computer, iPad, or android device for telehealth visits;
9. Negative urine pregnancy test at inclusion for females of reproductive potential (started the menstrual cycle);
10. For pediatric and adult females of reproductive potential (started the menstrual cycle): abstinence from sexual intercourse, or use of highly effective contraception for at least 30 days prior to screening, and agreement to use such a method during study participation and for three (3) days following the final topical system application;
11. For pediatric and adult males of reproductive potential: abstinence from sexual intercourse, or use of condoms or other methods to ensure effective contraception with partner during study participation and for three (3) days following the final topical system application; and
12. Able to read and speak English.

Exclusion Criteria:

1. Major soft tissue injury (fractures are only exclusionary if the injury is stabilized with a device, e.g., a hard cast, that cannot be removed to allow a topical system to be applied to the injured area);
2. Open skin lesion or any dermatological condition (e.g., skin infection, eczema) within the injured area;
3. Injury involves the spine, digits, hands, or bottom of foot;
4. Prior injury to the same site within the past 90 days;
5. Three or more other prior injuries (minor or major) to the region in the past;
6. Injury occurred more than 96 hours prior to study entry;
7. Prior use of topical medication to involved area within 48 hours of study entry;
8. Hypersensitivity disorders, including asthma or urticaria, but only if associated with exposure to aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) including diclofenac;
9. Coagulation defects;
10. Prior use of over the counter (OTC) analgesics or short-acting NSAIDs (ibuprofen, ketoprofen) within 6 hours of study entry (acetaminophen permitted up until the time of study entry);
11. Prior use of narcotic analgesics within seven (7) days of study entry;
12. Prior use of systemic anti-inflammatory steroidal drugs within 60 days of study entry;
13. Prior use of long-acting NSAIDs such as piroxicam or naproxen since injury;
14. Concomitant use of drugs which may be susceptible to interactions with diclofenac, or affect safety if used concomitantly (e.g., serotonin-selective reuptake inhibitors, lithium, digoxin, anticoagulants, antidiabetic agents, cyclosporin, methotrexate, quinolone antimicrobials, other NSAIDs, steroids and diuretics);
15. Participants with mental, behavioral, or neurodevelopmental disorders for which the relevant disorder(s) prevent compliance with the protocol;
16. Documented alcohol or drug abuse within 365 days of study entry;
17. Documented nicotine dependence within 365 days of study entry;
18. Current or prior history of severe cardiac, renal, or hepatic impairment or disease;
19. Severe systemic diseases (e.g., cancer, severe acute infection);
20. Any underlying disease or medication that severely compromises the participant's immune system;
21. Current or prior history of any chronic pain disorder;
22. Current or prior history of gastrointestinal bleeds or, ulcers;
23. Females who are pregnant or breast feeding; or
24. Participation in another clinical trial within 90 days of enrollment.

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Plasma diclofenac concentration of the Licart topical system as assessed by the Diclofenac pharmacokinetic profile. | 14-day treatment course
  Plasma diclofenac concentration, 24hours after initial topical system application (V2 and V5/EOS)
Local tolerability of the Licart topical system as assessed by a 7-point scale. | 14 days treatment course
  Local tolerability assessed via a 7-point scale by the PI or designee at V2, V3, V4 and V5/EOS. The 7-point scale is: Grade 0 = Absent Response with No Visible Change. Grade 1 = Vascular Dilation Stage Response with Visible Change of Faint Redness (not considered clinically relevant). Grade 2 = Vascular Dilation Stage Response with Visible Change of Moderate Redness. Grade 3 = Vascular Dilation Stage Response with Visible Change of Intense Redness. Grade 4 = Infiltration Stage Response with Visible Change of Redness with Edema or Papules. Grade 5 = Infiltration Stage Response with Visible Change of Redness with Weeping Vesicles, Blisters or Bullae. Grade 6 = Infiltration Stage Response with Visible Change of Redness with Extension of Effect Beyond Margin of Contact Site.
Adverse Events as assessed by the study team | 14 days treatment course
  Adverse Events for all participants as assessed by the study team during each visit throughout the duration of the study.
Pharmacokinetics of the Licart topical system as assessed by the activated partial thromboplastin time. | 14-day treatment course
  Plasma activated partial thromboplastin time (aPTT), 24hours after initial topical system application (V2 and V5/EOS).

SECONDARY OUTCOMES:
Analgesic Effect of the Licart topical system as assessed by the Wong-Baker FACES pain score assessment scale | 14-day treatment course
  Analgesic Effect of the Licart topical system as assessed by the Wong-Baker FACES pain score assessment scale every day (via participant's diary) and study visits on V2, V3, V4, V5/EOS. The pain score options are as followed: 0 = No Hurt, 2 = Hurts Little Big, 4 = Hurts Little More, 6 = Hurts Even More, 8 = Hurts Whole Lot, 10 = Hurts Worst. The lower the score, the better the outcome; the higher the score, the worse the outcome.
Global Response to Licart topical system as assessed by the Global Response to Therapy Investigator-reported questionnaire. | 14-day treatment course
  Global Response to Licart topical system as assessed by the Global Response to Therapy Investigator-reported questionnaire at V5/EOS.
Safety as assessed by vital signs - blood pressure. | 14 days treatment course
  Safety as assessed by vital signs - blood pressure (mm HG). Safety assessed by blood pressure (systolic and diastolic in mm HG) during each visit: V1, V2, V5/EOS.
Safety as assessed by vital signs - heart rate. | 14 days treatment course
  Safety assessed by heart rate (beats per minute) during each visit: V1, V2, V5/EOS.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Mautone, MD, Study Director — IBSA R&D Scientific Affairs
Locations (11):
- United States (11):
  - Applied Research Center, Little Rock, Arkansas
  - Atella Clinical Research, LLC., La Palma, California
  - University Clinical Research - Deland, LLC, DeLand, Florida
  - My Community Research, Inc., Miami, Florida
  - D & H Tamarac Research Centers, Inc., Tamarac, Florida
  - Research Integrity, Owensboro, Kentucky
  - Ascendant Research Clinic, LLC., Alamogordo, New Mexico
  - Prime Global Research Inc., The Bronx, New York
  - Ascendant Research Clinic, LLC., Marion, South Carolina
  - Next Level Urgent Care, Houston, Texas
  - AIM Trials, Plano, Texas

IPD SHARING:
Plan to Share IPD: No